CLINICAL TRIAL: NCT05115461
Title: Postural Stability in Patients With Lumbar Radiculopathy and it's Relation to Neuropathic Pain: a Cross Sectional Case-control Study
Brief Title: Neuropathic Pain and Postural Stability in Patients With Lumbar Radiculopathy
Status: Enrolling by invitation | Type: Observational
Sponsor: Bozyaka Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Buğra İnce, Assoc. Prof, Bozyaka Training and Research Hospital
Other Study IDs: 19663012TCS
Record Dates: First submitted 2021-11-01; First posted 2021-11-10 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Postural Stability; Balance; Distorted; Neuropathic Pain
MeSH Terms: conditions — Neuralgia | interventions — Surveys and Questionnaires; Equipment and Supplies; Restraint, Physical

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Radicular pain group: Patients presenting with lumbar radicular pain and MRI findings associated with radiculopathy
  Interventions: Device: Biodex Balance System™ SD; Other: questionnaires and inventories
- Control group: Age- and sex-matched control subjects without pain.
  Interventions: Device: Biodex Balance System™ SD

INTERVENTIONS:
Device: Biodex Balance System™ SD — Postural stability index values (anteroposterior, mediolateral and overall) will be measured for static and dynamic conditions.
Other: questionnaires and inventories — questionnaires and inventories related to primary end secondary outcomes will be applied and physical examination will be performed.
  Other Names: physical examination
  Groups: Radicular pain group

SUMMARY:
The aim of this study is to answer the questions below;

1. Is there a difference between patients with lumbar radiculopathy suffering from radicular pain and healthy subjects in terms of static and dynamic postural stability?
2. Is there a relationship between postural stability and the neuropathic characteristics of radicular pain?

DETAILED DESCRIPTION:
Patients presenting to our outpatient clinic with radicular pain and MRI findings associated with radiculopathy will be tested for static and dynamic postural stability. Patient demographics, pain intensity, neuropathic pain scores, and level of disability will also be recorded. The demographic data and postural stability scores will also be collected for the control subjects. Differences between the patient and control groups in terms of postural stability parameters will be sought. In addition, the relationship between the variables representing balance in the patient group and the neuropathic pain score and disability will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Having radicular pain due to lumbar disc herniation.
* Root compression on the dominant side on imaging.
* Root compression at no more than two levels.
* Radicular pain with at least 3 points on a numerical rating scale.

Exclusion Criteria:

* No radicular pain despite root compression on imaging.
* Midline disc herniation or root compression on the nondominant side.
* Radicular pain on the non-dominant side.
* Treatment with neuropathic pain medication or psychotropic medication.
* Loss of muscle strength on clinical examination.
* Evidence of lower extremity atrophy, joint contractures, shortening of limbs, or similar disabilities.
* Presence of vision loss, vestibular or neurological disorders that may cause balance disorders.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients presenting to our outpatient clinic with radicular pain and MRI findings associated with radiculopathy and age- and sex-matched healthy control subjects.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2021-11-10 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Dynamic Postural Stability | Once, at baseline
  Postural Stability Test will be performed via Biodex Balance System. This test assesses the patient's ability to maintain the center position (zero point) on a moving balance platform. The test protocol is performed with the following parameters: Duration: 20 seconds, Stability Level: 8, and Stance: two legs. Patients will complete a 1-minute pre-test trial to get used to the device. Then the test will be performed with 3 trials. The patient's performance will be noted as the overall stability index. A high stability index value indicates poor balance and stability.
Static Postural Stability | Once, at baseline
  Postural Stability Test will be performed via Biodex Balance System. This test assesses the patient's ability to maintain the center position (zero point) on a stable platform. The test protocol is performed with the following parameters: Duration: 20 seconds, Stability Level: Static, and Stance: both legs, alternating. Patients will complete a 1-minute pre-test trial to get used to the device. Then the test will be performed with 3 trials. The patient's performance will be noted as the overall stability index. A high stability index value indicates poor balance and stability.

SECONDARY OUTCOMES:
Neuropathic pain | Once, at baseline
  It will be assessed using the painDETECT questionnaire. The PainDETECT questionnaire contains nine questions, all based on self-assessment. Seven items are rated on a six-point Likert scale, ranging from 0-5. These seven questions query some sensations such as burning, tingling or prickling, allodynia, numbness, etc. Apart from these seven items, one item assesses the radiation of pain and another item asks about the temporal characteristics of pain. A total score of 12 or less indicates neuropathic component is unlikely, 13-18 means a possible neuropathic component and 19 or greater means that a neuropathic component is likely. In addition, there are three items in a separate section that measure the severity of pain at the time of assessment, on average, and at most in the last month. This section is not included in the assessment.
Disability | Once, at baseline
  It will be assessed using Quebec Back Pain Disability Scale. This scale contains 6 domains of activity affected by back pain: bed/rest (items 1-3), sitting/standing (items 4-6), ambulation (items 7-9), movement (items 10-12), bending/stooping (items 13-16), and handling of large/heavy objects (items 17-20). For each item, a 6-point Likert scale (0-5) to indicate the level of difficulty is used, where 0 = "not difficult at all," 1 = "minimally difficult," 2 = "somewhat difficult," 3 = "fairly difficult," 4 = "very difficult," and 5 = "unable to do." The total score is calculated by adding up the scores of each items. Scores range from 0 (no disability) to 100 (maximal disability).

CONTACTS AND LOCATIONS:
Overall Officials: Bugra Ince, MD, Principal Investigator — Bozyaka Training and Research Hospital; Taciser Kaya, Professor, Study Director — University of Health Sciences Izmır Faculty, Bozyaka Training and Research Hospital
Locations (1):
- Izmir Bozyaka Research and Training Hostpital, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lin SI, Lin RM. Sensorimotor and balance function in older adults with lumbar nerve root compression. Clin Orthop Relat Res. 2002 Jan;(394):146-53. doi: 10.1097/00003086-200201000-00017. PMID 11795726
- [Background] Kim KH, Leem MJ, Yi TI, Kim JS, Yoon SY. Balance Ability in Low Back Pain Patients With Lumbosacral Radiculopathy Evaluated With Tetrax: A Matched Case-Control Study. Ann Rehabil Med. 2020 Jun;44(3):195-202. doi: 10.5535/arm.19101. Epub 2020 May 29. PMID 32475097
- [Background] Sipko T, Kuczynski M. Intensity of chronic pain modifies postural control in low back patients. Eur J Pain. 2013 Apr;17(4):612-20. doi: 10.1002/j.1532-2149.2012.00226.x. PMID 23065907
- [Background] Tsigkanos C, Gaskell L, Smirniotou A, Tsigkanos G. Static and dynamic balance deficiencies in chronic low back pain. J Back Musculoskelet Rehabil. 2016 Nov 21;29(4):887-893. doi: 10.3233/BMR-160721. PMID 27341640
- [Background] Brech GC, Andrusaitis SF, Vitale GF, Greve JM. Correlation of disability and pain with postural balance among women with chronic low back pain. Clinics (Sao Paulo). 2012 Aug;67(8):959-62. doi: 10.6061/clinics/2012(08)17. No abstract available. PMID 22948466